CLINICAL TRIAL: NCT05146908
Title: Evaluation of Gastric Echography for Early Diagnosis of Nutritional Intolerance.
Acronym: NUTRIGUS 2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NGUYEN 2021-2
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Nutritional Intolerance
MeSH Terms: interventions — High-Energy Shock Waves; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in intensive care: Ventilated intubated patients for whom enteral nutrition is planned
  Interventions: Biological: 2 Blood samples from arterial and/or central venous catheters; Other: Echography; Other: Data collection

INTERVENTIONS:
Biological: 2 Blood samples from arterial and/or central venous catheters — 5 mL blood sample taken at the same time as a blood sample scheduled in regular patient management before the introduction of enteral nutrition and 24H after
Other: Echography — In 3 steps:
  * before initiation of enteral nutrition
  * 4h after initiation of enteral nutrition
  * After 24 hours of enteral nutrition
Other: Data collection — At inclusion:
  Calculation of severity scores; collection of reason for admission and demographic data; main comorbidities and treatments administered; the time between admission and nutritional recovery; risk factors for gastroparesis; current organ failure and supplements. Presence of parenteral nutrition, ongoing carbohydrate intake. Caloric objective.
  Within the first 24 hours, collection of:
  * echographic parameters at H0, H4 and H24
  * venous congestion parameters
  * biological parameters within 24 hours Constitution of a biobank (at H0 and H24)
  Within the first 7 days, collection of:
  * the occurrence or not of the primary endpoint (and time to occurrence).
  * symptoms of gastrointestinal dysfunction
  Within 30 days, collection of:
  * organ failure and replacement over the period, and mortality.
  * the occurrence or not of ventilator-associated lung disease (VAPD). Each patient is followed for 30 days. Survival will be assessed at 30 days before discharge from the study.

SUMMARY:
In intensive care, gastrointestinal dysfunction may occur in response to systemic insult. Acute gastrointestinal dysfunction (AGID) has been clinically defined by consensus and several grades of severity have been defined. Biomarkers of digestive distress have also been described in intensive care and can be measured directly in the plasma (lipopolysaccharide, intestinal fatty acid binding protein, citrulline, glucagon-like peptide-1).

Enteral nutrition is a frequent therapy in intensive care patients, and its administration is recommended. In general, nurtition is resumed early via a nasogastric tube in patients placed on mechanical ventilation. The resumption of nutrition can be seen as a "challenge" to the gastrointestinal tract, and may thus unmask underlying gastrointestinal dysfunction. Intolerance of enteral nutrition is a symptom of gastrointestinal dysfunction and is associated with poor clinical outcomes. Indeed, it is both a marker of severity by reflecting organ dysfunction and responsible for a reduction in caloric intake that can influence prognosis.

There is no consensus on the definition of intolerance to enteral nutrition. In practice, it is most often recognized because of regurgitation or vomiting, requiring reduction or discontinuation. In a recent review, the authors emphasize the need for digestive monitoring for early diagnosis of nutritional intolerance.

Gastric echography is a minimally invasive and reliable means of monitoring the gastric contents. In particular, the surface of the antrum has been validated as a way to diagnose a full stomach in intensive care. The measurement of echographic variations in gastric residue with the resumption of enteral nutrition could thus allow the early diagnosis of gastrointestinal dysfunction and food intolerance by preceding vomiting.

Our objective is to show the interest of echographic monitoring of the stomach during the resumption of enteral feeding for the diagnosis of nutritional intolerance. As nutritional intolerance is a symptom of gastrointestinal dysfunction, we will also study this phenomenon by measuring the associations between echographic data, clinical data and biomarkers of gastrointestinal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Next-of-kin/health care proxy has not objected to the inclusion of the patient
* Patient admitted to intensive care
* Predicted duration of MV > 48 hours
* Predicted start of enteral nutrition
* Time to the initiation of enteral nutrition and orotracheal intubation < 36 hours

Exclusion Criteria:

* Person subject to a measure of legal protection (curatorship, guardianship)
* Pregnant, parturient or breastfeeding women
* Minors
* Non echogenic patient or without an exploitable echographic window
* History of gastric or esophageal surgery
* Limitations of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU for whom enteral nutrition is planned
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Gastric antral surface in mm2 | Up to 24 hours of enteral nutrition
  Echographic measurement of the gastric antral area

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Derived] Berthoud V, Nguyen M, Vinay J, Perrot J, Pages PB, Guinot PG, Bouhemad B. Increase in Diaphragm and Expiratory respiratory muscles thickness is not associated with postoperative pulmonary complications after thoracic surgery: a prospective ultrasound cohort study. Anaesth Crit Care Pain Med. 2025 Nov 12:101683. doi: 10.1016/j.accpm.2025.101683. Online ahead of print. PMID 41238178